CLINICAL TRIAL: NCT00531505
Title: Morbid Obesity and Memory, Visceral and Subcutaneous mRNA Analysis, Body Composition, and Comorbidity Scale.
Brief Title: Obesity and Memory, mRNA, Body Composition, Comorbidity Scale
Acronym: 2a
Status: Terminated | Type: Observational
Why Stopped: Surgeon mistakenly removed liver and fat tissue from a non-LABS2a participant
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Bruce Wolfe, Professor of Surgery, Oregon Health and Science University
Other Study IDs: IRB00002571
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Obesity; Memory Deficits
Keywords: Obesity
MeSH Terms: conditions — Obesity; Memory Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver and fatty samples were voluntarily given by participant consent.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 2a: Morbid Obese individuals undergoing bariatric surgery (i.e. Laparoscopic Banding, Gastric Bypass). These individuals are a subset population of the greater Longitudinal Assessment of Bariatric Surgery (LABS-1) study population. This subpopulation engaged in memory tests as well as tissue extraction.

SUMMARY:
1. Briefly describe the purpose of this protocol. First purpose of the study is to understand the inheritance of morbid obesity.
2. Briefly summarize how participants are recruited. Volunteers will first learn of LABS-2a research opportunity at the Bariatric Surgery Informational meetings.
3. Briefly describe the procedures subjects will undergo.

   Participants will be asked to complete a set of memory tests. Fat and Liver samples will be removed during their weight loss surgery, specifically for this research study.
4. If applicable, briefly describe survey/interview instruments used. Memory tests will be performed to assess cognition.
5. Briefly describe how the data will be analyzed to address the purpose of the protocol.

The memory test data collected and compared against well established norms. Tissue samples will stored in a repository to be genetically studied for an indefinite amount of time. Genetic studies will be related to the disease of obesity and associated comorbidities brought on by the disease.

DETAILED DESCRIPTION:
1. Briefly describe the purpose of this protocol. First purpose of the study is to understand the inheritance of morbid obesity. If a gene or genes cause morbid obesity can be found, the diagnosis and treatment of morbid obesity may be improved. Second purpose is to learn more about the effects of weight loss on dementia, body composition, and comorbidity.
2. Briefly summarize how participants are recruited. Volunteers will first learn of LABS-2a research opportunity at the Bariatric Surgery Informational meetings. Subjects who express interest, will be screened through an IRB-approved informal telephone interview. If no exclusion criteria are identified, volunteers will be asked to provide IRB-approved consent. Recruitment will occur irrespective of race, religion or color.
3. Briefly describe the procedures subjects will undergo. Participants will be asked to complete a set of memory tests. These memory tests will be recorded on audio tape. BodPod will be used to measure their muscle, bone, and fat. The BodPod is an upright capsule that will enclose around a subject completely. BodPod uses the movement of air to measure muscle, and fat volumes. Participation in the memory testing portion and the BodPod portion of the research is optional. Fat and Liver samples will be removed during their weight loss surgery, specifically for this research study.
4. If applicable, briefly describe survey/interview instruments used. Memory tests will be performed to assess cognition. The Wechsler Memory Scale-Third Edition (WMS-III) and the Mini Memory State Examination (MMSE) will be the validated memory tests used. The WMS-III tests logical memory by having subjects recall short stories that were just read to them. The MMSE involves performing a set of requests that test orientation to time and place, immediate recall, short term verbal memory, calculation, language and construct ability.
5. Briefly describe how the data will be analyzed to address the purpose of the protocol.

The memory test data collected and compared against well established norms. Tissue samples will stored in a repository to be genetically studied for an indefinite amount of time. Genetic studies will be related to the disease of obesity and associated comorbidities brought on by the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age and undergo bariatric surgery by a LABS certified surgeon
* Previous enrollment in LABS-1 and LABS-2

Exclusion Criteria:

* Informed consent not obtained
* Prior bariatric surgery
* Unlikely to comply with follow-up protocol
* Unable to communicate with local study staff
* Extensive hearing impairment
* Medical conditions known to impact cognitive performance, including past or present history of traumatic brain injury or neurological disorder.
* Non-English speaking
* Inability to withhold caffeine and nicotine 2 hours before each visit, and alcohol 12 hours before each visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subset population of LABS-1 study population.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce M Wolfe, MD, Principal Investigator — Professor of Surgery, Oregon Health & Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States